CLINICAL TRIAL: NCT01895686
Title: Comparison of Visante and Cirrus Optical Coherent Tomography for Assessment of the Anterior Segment
Brief Title: Comparison of Gonioscopy With Cirrus and Visante
Acronym: ASOCT
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal Investigator, Wills Eye
Other Study IDs: 11-080E
Record Dates: First submitted 2012-12-20; First posted 2013-07-10 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2016-11

CONDITIONS: Open Angle Glaucoma; Narrow Angles; Angle Closure Glaucoma
Keywords: open angle glaucoma; narrow angles; angle closure glaucoma; gonioscopy; anterior segment OCT
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Open angle glaucoma: patients diagnosed with open angle glaucoma
- Narrow angle: patients diagnosed with narrow angles
- Angle Closure Glaucoma: patients diagnosed with angle closure glaucoma

SUMMARY:
The aim of this study is to analyze similarities and evaluate interchangeability of Visante and Cirrus OCT (optical coherent tomography)and to compare agreement between gonioscopy and the two systems for evaluation of anterior segment parameters.

DETAILED DESCRIPTION:
All participants underwent routine ophthalmic examination by their physician. Three independent examiners performed gonioscopy using Spaeth Gonioscopic Grading System. Findings were recorded independently along with risk assessment of angle being closed as: high, medium, and low or no risk. Patient information was not available to doctor during gonioscopy. One eye of each patient was imaged using both Visante and Cirrus OCT. Imaging was performed under scotopic and photopic conditions and obtained from horizontal (3:00 and 9:00 o'clock) and vertical (6:00 and 12:00 o'clock) meridians. The same experienced independent examiner performed all Cirrus measurements. Visante was performed by 3 trained technicians using same protocol.

OCT images were exported and masked to be evaluated for presence of open or closed anterior chamber angle. Masked images were presented with no other patient information available to two examiners with glaucoma training working together to score on basis of iridocorneal angle as, closed (0 degree), high possibility (10 degree), medium risk (20 degree), and low or no risk (> 30 degree).

ELIGIBILITY:
Inclusion Criteria:

• 18 years of age and older with open angle, narrow angle and angle closure

Exclusion Criteria:

• All lasers or intraocular surgery (cataract, glaucoma, retina, cornea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Phakic patients with open, narrow angle and angle closure glaucoma without prior intraocular surgery, including laser iridotomy or topical miotic use, were recruited for this study after Informed Consent was obtained.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
anterior angle measurement | 1 day
  comparison of AS assessment by Cirrus, Visante, gonioscopies

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Katz, MD, Principal Investigator — Glaucoma Service, Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Glaucoma Service, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Manuscript has been published in the Journal of Glaucoma.

REFERENCES:
- [Result] Hu CX, Mantravadi A, Zangalli C, Ali M, Faria BM, Richman J, Wizov SS, Razeghinejad MR, Moster MR, Katz LJ. Comparing Gonioscopy With Visante and Cirrus Optical Coherence Tomography for Anterior Chamber Angle Assessment in Glaucoma Patients. J Glaucoma. 2016 Feb;25(2):177-83. doi: 10.1097/IJG.0000000000000076. PMID 24844543